CLINICAL TRIAL: NCT01233141
Title: Phase IV Hospital Based Registry to Explore the Outcome of Chronic Critical Limb Ischemia
Brief Title: Viennese Registry on Patients With Chronic Critical Limb Ischemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Silvia Charwat, Medical University of Vienna
Other Study IDs: VICLI-2010
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2010-11

CONDITIONS: Chronic (> 2 Weeks) Critical Ischemia With Skin Defect in Lower Limbs
Keywords: peripheral artery disease stage IV (Fontaine's classification) or stage 5 and 6 (Rutherford's classification
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- one group only: all participants

SUMMARY:
The rationale of this study is to establish a registry to detect and follow patients with CLI treated in Vienna. The Vienna CLI registry is meant to document the incidence, prevalence, and actual outcome of CLI patients in a real world setting and should serve as a tool for the evaluation of medical, endovascular and surgical interventions. It will help determining the prognosis of individual patients and have impact on economic and political decisions in Vienna concerning this disease and the related costs.

DETAILED DESCRIPTION:
This is a prospective observational cohort study including consecutive patients with CLI. The study will be initiated as a single center evaluation and is intended to be step-wise expanded to a Vienna-wide systematic survey. The study will include patients with chronic critical limb ischemia and ischemic ulcerations as defined by Fontaine stage IV or Rutherford stages 5 & 6. The study will include all patients presenting with CLI to the participating centers including inpatients and outpatients.

Patients will be followed up 1 month, 3 months, 6 months, 12 months and then every 6 months. The study will be continued at least until the 5 year data of the last included patient are available.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (> 2 weeks) critical limb ischemia in one or both of the lower extremities with necrosis and/or gangrene in the limb (peripheral artery disease IV according to Fontaine's classification or Rutherford stage 5 & 6) of whatever genesis (atherosclerotic, aneurysmatic, embolic, inflammatory)
* ankle/brachial index < 0.4 or toe pressure < 30 mmHg
* Ability to give written informed consent

Exclusion Criteria:

* o Ulceration exclusively due to nonvascular causes like neuropathy (without coexisting hemodynamic impairment as defined above) or venous ulceration (without coexisting arterial impairment as defined above)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: tertiary care centre
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-01

PRIMARY OUTCOMES:
death | 5 years
ipsilateral amputation rate | 5 years
stroke | 5 years
myocardial infarction | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria